CLINICAL TRIAL: NCT02260752
Title: Comparing Options for Management: Patient Centered Results for Uterine Fibroids
Brief Title: Patient Centered Results for Uterine Fibroids
Acronym: COMPARE-UF
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00057883; RFA-HS-14-006 (Other Grant/Funding Number: Agency for Healthcare Research and Quality)
Record Dates: First submitted 2014-09-29; First posted 2014-10-09 (Estimated); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Fibroids, Uterine
MeSH Terms: conditions — Leiomyoma | interventions — Hysterectomy; Uterine Myomectomy; Nutrition Therapy; Endometrial Ablation Techniques; Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — blood assay
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Medical: Patients who receive medical therapy only for treatment of their uterine fibroids
  Interventions: Drug: Medical Therapy
- Procedure: Patients who have a hysterectomy, myomectomy, uterine arterial embolization, endometrial ablation, radiofrequency ablation, or magnetic resonance guided focused ultrasound to treat their UF.
  Interventions: Procedure: hysterectomy; Procedure: Uterine arterial embolization; Procedure: myomectomy; Procedure: endometrial ablation; Procedure: magnetic resonance guided focused ultrasound; Procedure: radiofrequency ablation

INTERVENTIONS:
Procedure: hysterectomy — surgical removal of the uterus
  Groups: Procedure
Procedure: Uterine arterial embolization — In uterine artery embolization, doctor uses a slender, flexible tube (catheter) to inject small particles (embolic agents) into the uterine arteries, which supply blood to your fibroids and uterus.the embolic agents are injected into these fibroid blood vessels. The goal is to block the fibroid vessels, starving the fibroids and causing them to shrink and die.
  Other Names: UAE
  Groups: Procedure
Procedure: myomectomy — surgical procedure to remove uterine fibroids, but does not remove uterus
  Groups: Procedure
Drug: Medical Therapy — treatment of uterine fibroids with only medications, no procedure or surgery is used
  Groups: Medical
Procedure: endometrial ablation — surgical procedure that destroys uterine lining via a telescope placed inside the uterus
  Other Names: NovaSure, Her Option, HydroTherm
  Groups: Procedure
Procedure: magnetic resonance guided focused ultrasound — procedure that destroys fibroids while inside an MRI machine
  Other Names: MRgFUS, ExAblate; Sonalleve
  Groups: Procedure
Procedure: radiofrequency ablation — procedure that uses heat to destroy uterine fibroids
  Other Names: Accessa
  Groups: Procedure

SUMMARY:
The overall goal of this project is to better enable patients with uterine fibroids (UF) to make informed decisions about treatment options by leveraging the highest possible evidence of healthcare quality. The foundation of this project will be a multi-site, prospective registry of a diverse group of women who have undergone either medical or surgical treatment for UF.

Specifically, the investigators are interested in: comparing management options for symptom relief; comparing management options for preserving reproductive function; and comparing effectiveness among different subpopulations, including consideration of patient needs and preferences of treatment options.

DETAILED DESCRIPTION:
COMPARE UF will enroll approximately 10,000 subjects across 9 clinical enrolling centers in the US. We anticipate recruitment to last approximately 24 months. Sites will consent interested patients and have them complete a patient contact information form to be used to contact the patient for telephone interviews. Following informed consent, the site will collect clinical information and several patient-reported outcomes scales, including the Uterine Fibroid Symptom Quality of Life Questionnaire (UFS-QOL), the Menopausal Rating Scale, and the EQ-5D, a standardized measure of general health outcomes.

In year 01 of this study, among patients receiving a procedure to treat their UF, 1000 will be asked to provide two blood samples: the first at time of enrollment (before the procedure) and the second at 12 months after the procedure. Samples will be evaluated for ovarian reserve via a blood assay measurement of anti-mullerian hormone.

Additionally, for patients who have a procedure to treat their UF, they will have a routine clinic follow-up visit, sometime between 6 - 12 weeks post procedure. Additional clinical data will be collected at this time.

For patients who are treated medically, there will be no further study-related clinic visits. Follow-up will occur exclusively by telephone.

All consented patients will complete telephone interviews at approximately 12, 24, and 36 months following the initial procedure. It is anticipated that patients enrolled during the first study year will complete a maximum of three years of follow-up. However, if additional funds become available, the investigators plan to extend the follow-up of enrolled patients to five years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of UF by imaging or pathology report within 2 years of enrollment initiation.
* Menstrual period within 12 months

Exclusion Criteria:

* Post-menopausal
* Men
* 55 years old or older

Ages: 18 Years to 54 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 10,000 patients diagnosed with UF between the ages of 18 and 54. Patients must have had a menstrual period within the last 12 months. Source documentation of UF must include either imaging or a pathology report.
Sampling Method: Non-Probability Sample
Enrollment: 3094 (Actual)
Dates: Start 2015-11; Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
change in symptom relief (patient interview) | 12, 24, 36 months
  degree to which bleeding and pain from uterine fibroids is alleviated

SECONDARY OUTCOMES:
change in preservation reproductive function (patient interview) | 12, 24, 36 months
  ability of a woman after receiving treatment for uterine fibroids can conceive and deliver a healthy baby

CONTACTS AND LOCATIONS:
Overall Officials: Evan R Myers, MD, Principal Investigator — Duke University
Locations (9):
- United States (9):
  - University of California Medical Centers, San Francisco, California
  - Uniformed Services University of the Health Sciences, Bethesda, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Inova Health Systems, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Anchan RM, Spies JB, Zhang S, Wojdyla D, Bortoletto P, Terry K, Disler E, Milne A, Gargiulo A, Petrozza J, Brook O, Srouji S, Morton CC, Greenberg J, Wegienka G, Stewart EA, Nicholson WK, Thomas L, Venable S, Laughlin-Tommaso S, Diamond MP, Maxwell GL, Marsh EE, Myers ER, Vines AI, Wise LA, Wallace K, Jacoby VL. Long-term health-related quality of life and symptom severity following hysterectomy, myomectomy, or uterine artery embolization for the treatment of symptomatic uterine fibroids. Am J Obstet Gynecol. 2023 Sep;229(3):275.e1-275.e17. doi: 10.1016/j.ajog.2023.05.020. Epub 2023 May 26. PMID 37244458
- [Derived] Anchan RM, Wojdyla D, Bortoletto P, Terry K, Disler E, Milne A, Gargiulo A, Petrozza J, Brook O, Srouji S, Morton CC, Greenberg J, Wegienka G, Stewart EA, Nicholson WK, Thomas L, Venable S, Laughlin-Tommaso S, Diamond MP, Maxwell GL, Marsh EE, Myers ER, Vines AI, Wise LA, Wallace K, Jacoby VL, Spies JB. A Comparative Analysis of Health-Related Quality of Life 1 Year Following Myomectomy or Uterine Artery Embolization: Findings from the COMPARE-UF Registry. J Womens Health (Larchmt). 2023 Apr;32(4):423-433. doi: 10.1089/jwh.2022.0133. Epub 2023 Jan 13. PMID 36637808
- [Derived] Wise LA, Thomas L, Anderson S, Baird DD, Anchan RM, Terry KL, Marsh EE, Wegienka G, Nicholson WK, Wallace K, Bigelow R, Spies J, Maxwell GL, Jacoby V, Myers ER, Stewart EA. Route of myomectomy and fertility: a prospective cohort study. Fertil Steril. 2022 May;117(5):1083-1093. doi: 10.1016/j.fertnstert.2022.01.013. Epub 2022 Feb 23. PMID 35216832
- [Derived] Wallace K, Stewart EA, Wise LA, Nicholson WK, Parry JP, Zhang S, Laughlin-Tommaso S, Jacoby V, Anchan RM, Diamond MP, Venable S, Shiflett A, Wegienka GR, Maxwell GL, Wojdyla D, Myers ER, Marsh E. Anxiety, Depression, and Quality of Life After Procedural Intervention for Uterine Fibroids. J Womens Health (Larchmt). 2022 Mar;31(3):415-424. doi: 10.1089/jwh.2020.8915. Epub 2021 Jun 8. PMID 34101502
- [Derived] Wegienka G, Stewart EA, Nicholson WK, Zhang S, Li F, Thomas L, Spies JB, Venable S, Laughlin-Tommaso S, Diamond MP, Anchan RM, Maxwell GL, Marsh EE, Myers ER, Vines AI, Wise LA, Wallace K, Jacoby VL. Black Women Are More Likely Than White Women to Schedule a Uterine-Sparing Treatment for Leiomyomas. J Womens Health (Larchmt). 2021 Mar;30(3):355-366. doi: 10.1089/jwh.2020.8634. Epub 2021 Feb 1. PMID 33524308
- [Derived] Laughlin-Tommaso SK, Lu D, Thomas L, Diamond MP, Wallace K, Wegienka G, Vines AI, Anchan RM, Wang T, Maxwell GL, Jacoby V, Marsh EE, Spies JB, Nicholson WK, Stewart EA, Myers ER. Short-term quality of life after myomectomy for uterine fibroids from the COMPARE-UF Fibroid Registry. Am J Obstet Gynecol. 2020 Apr;222(4):345.e1-345.e22. doi: 10.1016/j.ajog.2019.09.052. Epub 2019 Oct 31. PMID 31678093
- [Derived] Nicholson WK, Wegienka G, Zhang S, Wallace K, Stewart E, Laughlin-Tommaso S, Thomas L, Jacoby VL, Marsh EE, Wise L, Borah BJ, Spies J, Venable S, Anchan RM, Larry Maxwell G, Diamond M, Lytle B, Myers ER. Short-Term Health-Related Quality of Life After Hysterectomy Compared With Myomectomy for Symptomatic Leiomyomas. Obstet Gynecol. 2019 Aug;134(2):261-269. doi: 10.1097/AOG.0000000000003354. PMID 31306318
- [Derived] Stewart EA, Lytle BL, Thomas L, Wegienka GR, Jacoby V, Diamond MP, Nicholson WK, Anchan RM, Venable S, Wallace K, Marsh EE, Maxwell GL, Borah BJ, Catherino WH, Myers ER. The Comparing Options for Management: PAtient-centered REsults for Uterine Fibroids (COMPARE-UF) registry: rationale and design. Am J Obstet Gynecol. 2018 Jul;219(1):95.e1-95.e10. doi: 10.1016/j.ajog.2018.05.004. Epub 2018 May 8. PMID 29750955
- See also: COMPARE-UF Registry website — http://compare-uf.org/
- See also: Additional research study HSRP20194228 "Methods for the Design and Conduct of Subgroup Analysis in Observational Studies" — https://www.pcori.org/research-results/2019/developing-methods-comparing-outcomes-across-patient-groups-observational